CLINICAL TRIAL: NCT00776451
Title: Usability of the PreView PHP for Home Use in Intermediate Age Related Macular Degeneration Patients
Brief Title: Usability of the PreView PHP for Home Use in Intermediate AMD Patients
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Osnat Ehrman, Notal Vision
Organization: Notal Vision Inc. (Industry)
Other Study IDs: PHP-US-01
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Subjects diagnosed with Dry AMD

SUMMARY:
To demonstrate the ability of intermediate AMD subjects to follow the instructions for use and properly operate on their own the Preview PHP in home use environment, after going through training session.

DETAILED DESCRIPTION:
The study purpose is to demonstrate that the target population can use the system after going through a supervised training session. The PreView PHP will be operated in the same manner in the simulated setting as it will be in future home use.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study Subjects diagnosed as intermediate AMD in at least one eye
* Age ≥65 years
* VA with habitual correction better than 20/60 in the study eye
* Ability to speak, read and understand instructions in English or Hebrew
* Qualified to use the device by health care professional

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy, CFP.
* Any non-macular related ocular surgery or macular surgery performed within 3 months prior to study entry in the target eye
* Participation in another study with the exclusion of AREDS study
* Patients diagnosed with geographic atrophy (GA)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Dry AMD subjects
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who successfully completed the test by themselves, in a home simulated environment | 2 clinic visits

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bressler, Prof., Principal Investigator — JHMC
Locations (1):
- Belinson Medical Center, Petah Tikva, Israel

REFERENCES:
- See also: sponsor web site — http://www.notalvision.com